CLINICAL TRIAL: NCT01518556
Title: Phase I/II Clinical Study of Idarubicin Dose Intensification for Remission Induction Therapy in Acute Myeloid Leukemia Patients Age of 65 Years or Less
Brief Title: Safety and Efficacy Study of Idarubicin Dose Intensification to Treat Acute Myeloid Leukemia
Acronym: IDAML
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Konkuk University Medical Center (Other)
Collaborators: Chung-Ang University Hosptial, Chung-Ang University College of Medicine (Other); Seoul National University Hospital (Other); Ewha Womans University (Other); Samsung Medical Center (Other); Chonbuk National University Hospital (Other); Pusan National University Hospital (Other); Hanyang University Seoul Hospital (Other); Soon Chun Hyang University (Other)
Responsible Party: Principal Investigator, Mark Lee, Professor, Konkuk University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AML-2011-01
Record Dates: First submitted 2012-01-21; First posted 2012-01-26 (Estimated); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Leukemia, Myeloid, Acute
Keywords: Idarubicin; Remission Induction; Maximum Tolerated Dose; Survival
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Idarubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Idarubicin (Experimental): Idarubicin dose intensification for remission induction in acute myeloid leukemia
  Interventions: Drug: Idarubicin

INTERVENTIONS:
Drug: Idarubicin — In the phase I study, idarubicin dose is increased step by step as follows: 12 mg/m2/day for 3 days IV in the 1st step; 15 mg/m2/day for 3 days IV in the 2nd step; 18 mg/m2/day for 3 days IV in the 3rd step.
  In the phase II study, idarubicin dose is the maximum tolerated dose that is determined from the phase I study or 18 mg/m2/day for 3 days .
  Other Names: IDARU INJ

SUMMARY:
The purpose of this study is to determine whether idarubicin dose intensification is safe and effective as a remission induction therapy for acute myeloid leukemia.

DETAILED DESCRIPTION:
Up to nowadays, a standard induction therapy for acute myeloid leukemia(AML) has consisted of cytarabine 100-200 mg per square meter of body surface area(BSA) per day continuous infusion for 7 days with idarubicin 12 mg per square meter or daunorubicin 45 mg per square meter of BSA per day for 3 days. This standard therapy induces a complete remission(CR) in 50-75% of young adults and 40-50% of older adults. Recently two cooperative groups prospectively compared 45 mg per square meter of daunorubicin to 90 mg per square meter of BSA. They reported high-dose daunorubicin, as compared with a standard dose one, resulted in a significantly higher CR rate and improved overall survival(OS) up to age 65 without additional toxic effects.

Daunorubicin has been more commonly used anthracycline; however, idarubicin has a longer intracellular retention time and has shown more rapid clearance of marrow blasts. In the early 1990, three prospectively randomized studies showed that a combined regimen of idarubicin and cytarabine was superior to one of daunorubicin and cytarabine for the induction therapy of AML in adults. When they compared daunorubicin 45-50 mg per square meter with idarubicin 12-13 mg per square meter for induction therapy, there were no significant differences in hematologic and non-hematologic toxicities, including cardiac toxicity.

Phase I studies of idarubicin in patients with acute leukemia and chronic myelogenous leukemia in blast crisis reported the dose-limiting toxicities(DLT) were stomatitis and anorexia at the maximum tolerated dose(MTD) of 15 mg per square meter of BSA per day for 3 days. Based on the results of these studies, the investigators have generally administered idarubicin 12 mg per square meter per day for 3 days for the remission induction therapy of AML. Meanwhile Sanz et al. had administered idarubicin 12 mg per square meter per day for 4 days in patients with acute promyelocytic leukemia, and Tedeschi et al. had done a single high-dose idarubicin 40 mg per square meter combined with high-dose cytarabine 3 g per square meter per day for 5 days in patients with acute lymphoblastic leukemia, with no significant increase of severe toxicity. The MTD of idarubicin should be reevaluated in the treatment of acute leukemia, especially in the era of granulocyte colony-stimulating factor and better supportive care available.

In this phase I study, idarubicin 12 mg per square meter of BSA per day for 3 days will be given to three patients at the first stage and then the idarubicin dose will be increased by 3 mg per square meter of BSA each stage. The phase I study consists of 3 stages and the idarubicin dose will be increased up to 18 mg per square meter of BSA per day for 3 days unless DLTs do not develop in more than 33% of enrolled patients at each stage. In the subsequent phase II study, the MTD being determined from the phase I study or 18 mg per square meter of idarubicin will be given to the enrolled patients. There were three large studies which enrolled a total of 942 previously untreated adult patients with AML and in which idarubicin 12-13 mg per square meter of BSA per day for 3 days and cytarabine 100 mg per square meter daily for 7 days were administered intravenously. Therefore, the investigators can adopt them as historical control groups in terms of statistical assessment.

In conclusion, the investigators desire to determine the safety and effectiveness of the intensified dose of idarubicin in the treatment of acute myeloid leukemia through this phase I and II study.

ELIGIBILITY:
Inclusion Criteria:

* Patient has been fully informed, has complete understanding fo this study, and has given voluntary written informed consent to comply with the protocol requirements.
* previously untreated de novo or secondary acute myeloid leukemia, including biphenotypic leukemia
* age between 20 and 65 years
* adequate organ functions, unless these abnormalities are attributable to leukemia
* left ventricular ejection fraction > 45%
* serum creatinine < 1.5 x upper limit of normal
* total bilirubin < 1.5 x upper limit of normal
* alanine transferase and aspartate transferase < 2.5 x upper limit of normal if liver function abnormality is attributable to underlying leukemia, ALT and AST < 5 x upper limit of normal
* Eastern Cooperative Oncology Group performance status score of 0 to 2

Exclusion Criteria:

* hypersensitivity to the study drug
* any other malignancies within 3 years, except for cured non-melanoma skin cancer and curatively treated in situ carcinoma of the cervix
* New York Heart Association class III or IV heart failure, severe uncontrolled cardiac disease or myocardial infarction within the previous 6 months prior to the date of consent
* incapable of giving voluntary written informed consent to comply with the protocol requirements, which results from drug or alcohol intoxication, or neurological or psychiatric disorders
* pregnant or breastfeeding
* recent chemotherapy within 4 weeks prior to this study treatment
* acute promyelocytic leukemia
* current or recent treatment with any other investigational medicinal product within 28 days prior to this study enrollment
* unsuitable for this study, in the investigator's opinion

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2011-07 (Actual); Primary Completion 2025-03 (Actual); Study Completion 2025-03 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose of idarubicin in the phase I study. | Within 2 months after induction therapy in the phase I study.
  The study design is adopted from traditional 3+3 design for phase I cancer clinical trials. The first three patients are treated at a starting dose (level 1). If none of the three patients experiences a DLT(dose-limiting toxicity), another group of three patients will be treated at the next higher dose level. However, if one of the first three patients experiences a DLT, three more patients will be treated at the same dose level. The dose increment continues until at least two patients among a cohort of three to six patients experience DLTs.The maximum tolerated dose is defined as the dose level just below this toxic dose level.
Complete remission rate in the phase II study. | Within 2 months after induction therapy therappy in the phase II study.
  A complete remission designation requires that the patient achieve the morphologic leukemia-free state and have an absolute neutrophil count of more than 1000 per microliter and platelets of more than 100000 per microliter. Hemoglobin concentration or hematocrit has no bearing on remission status, although the patient must be independent of transfusions.

SECONDARY OUTCOMES:
Dose-limiting toxicity in the phase I study. | Within 2 months after induction therapy in the phase I study.
  Hematologic dose limiting toxicities (DLTs) are defined as the time to recovery of neutrophils (absolute neutrophil count of more than 500 per microliter) or platelets (platelet count of more than 20000 per microliter) exceeding 42 days after the start of induction therapy. Non-hematologic DLTs are defined as grade 4 or 5 toxicities.
Event-free survival and overall survival in the phase II study. | Within 5 years after induction therapy in the phase II study.
  Event-free survival is defined for all patients and measured from the date of entry on study. It is measured until treatment failure, relapse from CR, or death from any cause, whichever occurs first. Overall survival is defined for all patients in a trial, and measured from the date of entry onto a study until death from any cause. For a patient who is not known to have died by the end of study follow-up, observation of OS is censored on the date he or she was last known to be alive.

CONTACTS AND LOCATIONS:
Overall Officials: Mark H Lee, M.D., Ph.D., Principal Investigator — Konkuk University Medical Center
Locations (1):
- Division of Hematology-Oncology, Konkuk University Medical Center, Seoul, South Korea